CLINICAL TRIAL: NCT04224155
Title: A Prospective, Multicenter, Randomized, Masked, Controlled Clinical Study to Evaluate the Safety and Performance of the enVista® One-Piece Hydrophobic Acrylic Trifocal Intraocular Lens in Subjects Undergoing Cataract Extraction
Brief Title: Clinical Study to Evaluate the Safety and Performance of the enVista® One-Piece Hydrophobic Acrylic Trifocal Intraocular Lens in Subjects Undergoing Cataract Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 900
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- enVista MX60EFH trifocal intraocular lens (IOL) (Experimental)
  Interventions: Device: enVista MX60EFH trifocal intraocular lenses (IOLs)
- enVista MX60E monofocal intraocular lens (IOL) (Active Comparator)
  Interventions: Device: enVista MX60E monofocal intraocular lenses (IOLs)

INTERVENTIONS:
Device: enVista MX60EFH trifocal intraocular lenses (IOLs) — enVista MX60EFH trifocal intraocular lenses (IOLs) implanted bilaterally
  Arms: enVista MX60EFH trifocal intraocular lens (IOL)
Device: enVista MX60E monofocal intraocular lenses (IOLs) — enVista MX60E monofocal intraocular lenses (IOLs) implanted bilaterally
  Arms: enVista MX60E monofocal intraocular lens (IOL)

SUMMARY:
The objective of the study is to evaluate the safety and performance of the enVista trifocal intraocular lens when implanted in the capsular bag.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older on the date the Informed Consent Form (ICF) is signed.
* Subjects must have the capability to understand and provide written informed consent on the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved Informed Consent Form (ICF) and authorization as appropriate for local privacy regulations.
* Subjects must have a Best-corrected Distance Visual Acuity (CDVA) equal to or worse than 20/40 in at least one eye, with or without a glare source, due to a clinically significant cataract (cortical, nuclear, subcapsular, or combination) that is considered amenable to treatment with standard phacoemulsification cataract extraction and capsular IOL implantation.
* Subjects must have a Best-corrected Distance Visual Acuity (CDVA) projected to be equal to or better than 20/32 after IOL implantation in each eye, as determined by the medical judgment of the Investigator or measured by potential acuity meter (PAM) testing, if necessary.
* Subjects must have clear intraocular media other than the cataract in both eyes.
* Subjects must have discontinued use of contact lenses for at least 2 weeks (for hard lenses) or 3 days (for soft lenses) prior to the pre-operative examination and must be willing to refrain from use of contact lenses throughout the clinical study.
* Contact lens wearers must demonstrate a stable refraction (within ±0.50 D for both sphere and cylinder) in both eyes, as determined by distance manifest refraction on two consecutive examination dates after discontinuation of contact lens wear.
* Subjects must require an IOL power from +16.0 diopter (D) to +27.0 D in both eyes.
* Subjects must be willing and able to comply with all treatment and follow-up study visits and procedures, and to undergo second eye surgery within 7-30 days of the first eye surgery.

Exclusion Criteria:

* Subjects who have participated in an investigational drug or device clinical investigation within 30 days prior to entry into this study and/or will participate in another investigation during the period of study participation.
* Subjects who have any corneal pathology (e.g., significant scarring, guttata, inflammation, edema, dystrophy, etc.) in either eye. . '
* Subjects who have significant anterior segment pathology that might increase intraoperative risk or compromise IOL stability (e.g., pseudoexfoliation syndrome, synechiae, iris atrophy, traumatic cataract, lens subluxation, traumatic zonulolysis, zonular dialysis, evident zonular weakness or dehiscence, hypermature or brunescent cataract, etc.) in either eye.
* Subjects who have uncontrolled glaucoma in either eye.
* Subjects who have previous retinal detachment or clinically significant retinal pathology involving the macula in either eye.
* Subjects who have proliferative or non-proliferative diabetic retinopathy in either eye.
* Subjects who have a congenital ocular anomaly (e.g., aniridia, congenital cataract) in either eye.
* Subjects with instability of keratometry or biometry measurements.
* Subjects using any systemic or topical drug known to interfere with visual performance, pupil dilation, or iris structure within 30 days of enrollment or during the study.
* Subjects who have current or previous usage of an alpha-I-selective adrenoceptor blocking agent or an antagonist of alpha IA adrenoceptor (e.g., Flomax® (tamsulosin HCI), Terazosin, or Cardura).
* Subjects who have a history of chronic or recurrent inflammatory eye disease (e.g., iritis, scleritis, iridocyclitis, or rubeosis iridis) in either eye.
* Subjects who have a visual disorder, other than cataracts, that could potentially cause future acuity losses to a level of 20/ I 00 or worse in either eye.
* Subjects who have had previous intraocular or corneal surgery in either eye, with the exception of laser trabeculoplasty.
* Subjects with any preoperative infectious conjunctivitis, keratitis, or uveitis in either eye.
* Subjects who have a preoperative corneal astigmatism> 1.0 D in either eye as measured by corneal topography, irregular astigmatism, or skewed radial axis (note: corneal incisions intended specifically to reduce astigmatism are not allowed during the study).
* Subjects who cannot achieve a minimum pharmacologic pupil dilation of 5.0 mm in both eyes.
* Subjects who may be expected to require a combined or other secondary surgical procedure in either eye.
* Females of childbearing potential (those who are not surgically sterilized or at least 12 months postmenopausal) are excluded from enrollment in the study if they are nursing, lactating, currently pregnant or plan to become pregnant during the study. Females of childbearing potential must be willing to practice effective contraception for the duration of the study.
* Subjects with any other serious ocular pathology or underlying systemic medical condition (e.g., uncontrolled diabetes) or circumstance that, based on the Investigator's judgment, poses a concern for the subjects' safety or could confound the results of the study.
* Subjects with abnormal pupillary dilation dynamics (as determined by the medical judgment of the investigator) or eccentric or ectopic pupils in either eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch & Lomb Incorporated
Locations (9):
- Canada (9):
  - Bausch Site 106, Calgary, Alberta
  - Bausch Site 102, Concord, Ontario
  - Bausch Site 103, Mississauga, Ontario
  - Bausch Site 105, Toronto, Ontario
  - Bausch Site 107, Toronto, Ontario
  - Bausch Site 108, Vaughan, Ontario
  - Bausch Site 101, Boisbriand, Quebec
  - Bausch Site 113, Longueuil, Quebec
  - Bausch Site 104, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Muzychuk A, Harasymowycz P. Efficacy and safety evaluation of a new full visual range vs monofocal intraocular lens in patients with cataract: randomized, controlled Canadian clinical trial. J Cataract Refract Surg. 2025 Oct 1;51(10):867-875. doi: 10.1097/j.jcrs.0000000000001714. PMID 40490939

RESULTS

PARTICIPANT FLOW:
Groups:
- enVista MX60EFH Trifocal Intraocular Lens (IOL): Subjects assigned to enVista MX60EFH trifocal intraocular lenses (IOLs)
- enVista MX60E Monofocal Intraocular Lens (IOL): Subjects assigned to enVista MX60E monofocal intraocular lenses (IOLs)
Period: Overall Study
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
Started | 111 | 54
Completed | 110 | 52
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL) | Total
Number analyzed (Participants) | 111 | 54 | 165
Number analyzed (Eyes) | 222 | 107 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (7.66) | 66.8 (7.77) | 67.7 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 27 | 82
  Male | 56 | 27 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 106 | 53 | 159
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 11 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 80 | 40 | 120
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 111 | 54 | 165

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: All serious adverse events through Post-Operative Visit 4 (Day 120 to Day 180 after second eye IOL implantation)
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Measure: Count of Participants; unit: Participants
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
Number analyzed (Participants) | 111 | 54
Participants
  Diverticulitis | 1 | 0
  Neck pain | 1 | 0
  Neoplasm malignant | 1 | 0
  Cerebrovascular accident | 0 | 1
  Dry age-related macular degeneration | 1 | 0

2. Primary Outcome: Cumulative Rate of Secondary Surgical Interventions Due to the Optical Properties of the Lens
Description: The cumulative rate of secondary surgical interventions (SSI) due to the optical properties of the lens, through Post-Operative Visit 4 (Day 120 to Day 180 after second eye IOL implantation). The rate was determined as the number of eyes with an SSI related to the optical properties of the IOL divided by the total number of eyes.
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
Number analyzed (Participants) | 111 | 54
Number analyzed (Eyes) | 222 | 107
Eyes | 0 | 0

3. Primary Outcome: Photopic Uncorrected Distance Visual Acuity (UDVA) for First Implanted Eyes
Description: Photopic uncorrected distance visual acuity (UDVA) for first implanted eyes at 4 m at Post.Operative Visit 4 (Day 120 to Day 180 after second eye IOL implantation)
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Population: Per Protocol Set
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
Number analyzed (Participants) | 108 | 50
logMAR | 0.121 (0.1343) | 0.044 (0.1224)

4. Primary Outcome: Photopic Uncorrected Near and Intermediate Visual Acuity (UNVA and UIVA) for First Implanted Eyes at 40 cm and 66 cm, Respectively
Description: Photopic uncorrected near and intermediate visual acuity (UNVA and UIVA) for first implanted eyes at 40 cm and 66 cm, respectively, at Post-Operative Visit 4 (Day 120 to Day 180 after second eye IOL implantation)
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
Number analyzed (Participants) | 111 | 54
logMAR
  UNVA | 0.210 (0.1294) | 0.476 (0.1587)
  UIVA | 0.163 (0.1247) | 0.286 (0.1543)

5. Primary Outcome: The Incidence of Adverse Events (AEs), Through Postoperative Visit 4 (Day 120 to Day 180 After Second Eye IOL Implantation), Compared to ISO Safety and Performance Endpoint Rates.
Description: The incidence of adverse events (AEs), through Postoperative Visit 4 (Day 120 to Day 180 after second eye IOL implantation), compared to ISO Safety and Performance Endpoint rates as defined in ISO 11979-7:2018 and EN ISO 11979-7:2018 Annex E. The observed AE rate was calculated as 100 multiplied by the number of eyes with the specific treatment-emergent event divided by the number of implanted eyes.
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL)
Number analyzed (Participants) | 111
Number analyzed (Eyes) | 222
Eyes
  Cystoid macular oedema | 3
  Hypopyon | 0
  Endophthalmitis | 0
  Lens dislocated from posterior chamber | 0
  Pupillary block | 0
  Retinal detachment | 0
  SSI | 0

6. Secondary Outcome: Incidence of Subjects Experiencing at Least One Severe Visual Disturbance
Description: The incidence of Patient-Reported Outcomes Set subjects experiencing at least one severe visual disturbance, defined as the highest grade of severity or bothersomeness (separately) reported by subjects using the Quality of Vision (QoV) questionnaire at Post-Operative Visit 4 (Day 120 to Day 180 after second eye IOL implantation). Incidence was calculated as 100 multiplied by Count of Participants experiencing at least one severe visual disturbance divided by Number of Participants Analyzed.
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Population: PRO Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
Number analyzed (Participants) | 110 | 52
Participants | 16 | 4

7. Secondary Outcome: Photopic Contrast Sensitivity With Glare at Post-Operative Visit 4
Description: Photopic contrast sensitivity with glare at Post-Operative Visit 4 (Day 120 to Day 180 after second eye IOL implantation).
  Binocular photopic (approximately 85 cd/m2) contrast sensitivity with glare was tested at spatial frequencies of 3, 6, 12 and 18 cycles per degree (cpd) and was assessed in log units.
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Measure: Mean (Standard Deviation); unit: log value
Units Other Than Participants: eyes
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
Number analyzed (Participants) | 64 | 18
Number analyzed (eyes) | 64 | 18
log value
  At 3 cpd | 1.703 (0.3497) | 1.965 (0.3259)
  At 6 cpd | 1.544 (0.2989) | 1.894 (0.3325)
  At 12 cpd | 1.249 (0.3330) | 1.366 (0.3475)
  At 18 cpd | 0.749 (0.3483) | 1.016 (0.3203)

8. Secondary Outcome: Mesopic Contrast Sensitivity With Glare at Post-Operative Visit 4
Description: Mesopic contrast sensitivity with glare at Post-Operative Visit 4 (Day 120 to Day 180 after second eye IOL implantation). Binocular mesopic (2.5 to 3.2 cd/m2) contrast sensitivity with glare was tested at spatial frequencies of 1.5, 3, 6 and 12 cpd and was assessed in log units.
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Measure: Mean (Standard Deviation); unit: log value
Units Other Than Participants: eyes
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
Number analyzed (Participants) | 64 | 18
Number analyzed (eyes) | 64 | 18
log value
  At 1.5 cpd | 1.534 (0.3585) | 1.701 (0.3113)
  At 3 cpd | 1.552 (0.3405) | 1.884 (0.2853)
  At 6 cpd | 1.188 (0.3020) | 1.577 (0.2668)
  At 12 cpd | 0.605 (0.3235) | 0.882 (0.2936)

9. Secondary Outcome: Mesopic Contrast Sensitivity Without Glare at Post-Operative Visit 4
Description: Mesopic contrast sensitivity without glare at Post-Operative Visit 4 (Day 120 to Day 180 after second eye IOL implantation). Binocular mesopic (2.5 to 3.2 cd/m2) contrast sensitivity without glare was tested at spatial frequencies of 1.5, 3, 6 and 12 cpd and was assessed in log units.
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Measure: Mean (Standard Deviation); unit: log value
Units Other Than Participants: eyes
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
Number analyzed (Participants) | 64 | 18
Number analyzed (eyes) | 64 | 18
log value
  At 1.5 cpd | 2.024 (0.2661) | 1.943 (0.4097)
  At 3 cpd | 1.999 (0.2995) | 2.100 (0.3775)
  At 6 cpd | 1.574 (0.3156) | 1.753 (0.4634)
  At 12 cpd | 0.881 (0.3646) | 1.014 (0.3298)

10. Secondary Outcome: IOL Rotation for All Eyes at Post-Operative Visit 4
Description: IOL rotation for all eyes at Post-Operative Visit 4 (Day 120 to Day 180 after second eye IOL implantation)
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Eyes
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL)
Number analyzed (Participants) | 111
Number analyzed (Eyes) | 222
degrees | 2.21 (2.501)

11. Secondary Outcome: Change From Baseline ( Preoperative ) in Uncorrected Photopic Near and Intermediate Visual Acuity (UNVA and UIVA) at 40 cm and 66 cm, Respectively, for First Implanted Eyes to Post-Operative Visit 4
Description: Change from baseline ( preoperative ) in uncorrected photopic near and intermediate visual acuity (UNVA and UIVA) at 40 cm and 66 cm, respectively, for first implanted eyes to Post-Operative Visit 4 (Day 120 to Day 180 after second eye IOL implantation)
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
Number analyzed (Participants) | 111 | 54
logMAR
  UNVA | -0.502 (0.2947) | -0.157 (0.3062)
  UIVA | -0.505 (0.2983) | -0.305 (0.3216)

ADVERSE EVENTS:
Time Frame: Day 120 to Day 180 after second eye IOL implantation
Description: Ocular Adverse Events
Groups:
- enVista MX60EFH Trifocal Intraocular Lens (IOL): Subjects implanted with enVista MX60EFH trifocal intraocular lenses (IOLs). For ocular AEs, the number of eyes at risk were 222 for the enVista MX60EFH trifocal intraocular lens (IOL) group.
- enVista MX60E Monofocal Intraocular Lens (IOL): Subjects implanted with enVista MX60E monofocal intraocular lenses (IOLs). For ocular AEs, the number of eyes at risk were 107 for the enVista MX60E monofocal intraocular lens (IOL) group.
Arm/Group | enVista MX60EFH Trifocal Intraocular Lens (IOL) | enVista MX60E Monofocal Intraocular Lens (IOL)
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/54
Serious Adverse Events (participants affected / at risk) | 4/111 | 1/54
Other Adverse Events (participants affected / at risk) | 21/111 | 8/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | enVista MX60EFH Trifocal Intraocular Lens (IOL) (N=111) | enVista MX60E Monofocal Intraocular Lens (IOL) (N=54)
Dry age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | enVista MX60EFH Trifocal Intraocular Lens (IOL) (N=111) | enVista MX60E Monofocal Intraocular Lens (IOL) (N=54)
Punctate keratitis (Eye disorders) | 21 (29) | 8 (10)
Visual Acuity Reduced (Eye disorders) | 2 (2) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact Sponsor directly for details

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT04224155/Prot_SAP_000.pdf